CLINICAL TRIAL: NCT07116486
Title: Phase 1, Single-site, Single-arm, Clinical Imaging, and Blood-based Biomarker Trial Utilizing 18F-FSPG PET to Guide Therapy in Hepatocellular Carcinoma
Brief Title: A Trial Utilizing 18F-FS PG PET to Guide Therapy in Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1073; NCI-2025-06275 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-08-07; First posted 2025-08-11 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Participants will be scheduled for a baseline investigational 18F-FSPG PET/CT scan within 4 weeks of SOC CT and no more than 2 weeks prior to Y90 treatment.
  Interventions: Diagnostic Test: Radiopharmaceutical 18F-FSPG

INTERVENTIONS:
Diagnostic Test: Radiopharmaceutical 18F-FSPG — Given by injection

SUMMARY:
To evaluate the relationship between 18F-FSPG uptake in HCC lesions, ctDNA in blood and clinical response to Y90 radioembolization therapy in patients with hepatocellular carcinoma (HCC) by SOC imaging.

DETAILED DESCRIPTION:
Primary Objectives:

1. To establish whether pre-treatment 18F-FSPG can be utilized as an imaging marker to predict response/resistance to Y90 treatment,
2. To determine whether there is a correlation between change in 18F-FSPG uptake in HCC lesions and change in levels of ctDNA in the blood prior to and post-Y90 radioembolization and response to treatment as assessed by SOC imaging at 3-, 6-, 9-, and 12-months following the procedure.

Secondary Objectives:

1. To determine if 18F-FSPG PET can visualize residual disease,
2. To determine if ctDNA can detect residual disease,
3. To determine the concordance of tumor detection by 18F-FSPG PET/CT imaging and SOC imaging.
4. To establish whether 18F-FSPG uptake and levels of ctDNA can be utilized as imaging and bloodbased markers, respectively, to inform the response to therapy or lack thereof earlier than SOC imaging.
5. To evaluate the relationship between 18F-FSPG PET, ctDNA, and SOC imaging to TTP or PFS.
6. To evaluate voxel-wise relationships between 18F-FSPG intra-tumoral accumulation and SOC imaging.
7. To evaluate the treatment response using the mRECIST and LI-RADS criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of HCC with one or more of the following:

   1. Liver mass with non-rim arterial phase hyperenhancement (APHE) and one of the following:

      1. 10-19 mm with ≥ 2 additional major features according to LI-RADS criteria ("washout", enhancing "capsule", and/or threshold growth),
      2. 10-19 mm with "washout" and visibility at antecedent ultrasound (US) but with no "capsule" or threshold growth,
      3. 10-19 mm with ≥50% size increase in ≤6 months but with no "washout" or "capsule" or
      4. ≥20 mm with ≥1 additional major feature according to LI-RADS criteria ("washout", enhancing "capsule", or threshold growth).
   2. Lesions that meet LI-RADS 4 criteria or
   3. Lesions that meet LI-RADS 5 criteria or
   4. Suggestive imaging findings plus Alpha Fetoprotein (AFP) > 200 mg/dL or
   5. Tumor confirmed by arteriography or
   6. Pathologic confirmation of tumor and
2. Patients with HCC must be a candidate for Y90 radioembolization monotherapy. and
3. Each patient must have completed conventional imaging and staging and CT before initiation of the investigational PET studies.
4. Age ≥18 years. Because no dosing or adverse event data are currently available on the use of 18F-FSPG in patients <18 years of age, children are excluded from this study.
5. The effects of 18F-FSPG on the developing human fetus are unknown. For this reason women and men of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

   * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
   * History of hysterectomy or bilateral salpingo-oophorectomy.
   * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
   * History of bilateral tubal ligation or another surgical sterilization procedure.

     * Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
     * Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of 18F-FSPG administration.
6. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Patients under the age of 18 will be excluded from the this study.
2. Patients who have HCC but are not candidates for Y90 radioembolization monotherapy.
3. Pregnant and breastfeeding patients. Pregnant women are excluded from this study because 18F-FSPG as a radiotracer has a potential teratogenic or abortifacient effect. Because there is an unknown but potential risk for adverse events in nursing infants secondary to administration of the tracer 18F-FSPG to the mother, breastfeeding should be discontinued.
4. Patients with poorly controlled diabetes mellitus (fasting blood glucose level > 200 mg/dL).
5. Patients with psychiatric illness/social situations that would limit compliance with study requirements.
6. Patients who have not recovered from AEs or had allergic reactions to similar compounds should be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Simone Krebs, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org